CLINICAL TRIAL: NCT05253092
Title: The Effect of Mindfulness Meditation on Sleep Quality and Perceived Stress of Students in Higher Education
Brief Title: The Effects of Mindfulness Meditation on Sleep Quality and Perceived Stress
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of the Sciences in Philadelphia (Other)
Responsible Party: Principal Investigator, Nabila Enam, Assistant Professor, University of the Sciences in Philadelphia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1519081-3
Record Dates: First submitted 2022-02-01; First posted 2022-02-23 (Actual); Last update posted 2022-08-29 (Actual); Status verified 2022-08

CONDITIONS: Sleep
Keywords: Sleep, perceived stress, higher education, mindfulness meditation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Virtual mindfulness meditation (Other)
  Interventions: Other: Virtual mindfulness meditation

INTERVENTIONS:
Other: Virtual mindfulness meditation — Subjects will participate in 30 minutes of a virtual mindfulness meditation session, totaling eight sessions.

SUMMARY:
Higher education students 18 years or older will participate in 8- virtual mindfulness meditation sessions over 3 to 4 weeks (minimum of 3 sessions per week). Each session will be 30 minutes long, 15 minutes for guided mindfulness meditation run by researchers, followed by a short discussion period to understand mindfulness meditation better. Before starting the mindfulness meditation session, baseline data will be collected.

DETAILED DESCRIPTION:
Sleep consider a restorative occupation that affects other daily activities, such as academic performance. Mindfulness meditation may improve sleep quality and decrease perceived stress in higher education students. There is limited research on virtual mindfulness meditation involving sleep quality and perceived stress in higher education students. The researchers will measure changes in sleep quality and perceived stress after participants completed 8- virtual mindfulness meditation sessions using PSQI, PSS, and the Fitbit Inspire 2™.

ELIGIBILITY:
Inclusion Criteria:

* Must be a student at the University of the Sciences
* 18 years or older and fluent in English
* Students must have access to a device with internet connection and Zoom capabilities
* Students must have a smartphone to download the Fitbit®: Health & Wellness application.

Exclusion Criteria:

* Students who do not attend the University of the Sciences
* Students do not have access to an internet connection and an electronic device
* Students do not comprehend and speak English
* Students under the age of 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-01-17 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
Pittsburgh Sleep Quality Index (PSQI) | 10 minutes
  The PSQI is a nine-question, self-report index that assesses quality of sleep. The questionnaire is made up of scaled responses from 0-3; 0 is not during the past month, 1 is less than once a week, 2 is once or twice a week, and 3 is three or more times a week. If the individual scores higher than a 5 overall, it is an indication of poor sleep quality.

SECONDARY OUTCOMES:
Perceived Stress Scale (PSS) | 10 minutes
  The PSS is a self-report, ten question scale that measures perceived stress. This assessment uses a five-point Likert type scale to record responses. Responses range from 0, indicating "never" to 4, indicating "very often". A higher total score indicates higher perceived stress. Questions are general and ask about stressors in the last month.

OTHER OUTCOMES:
Fitbit Inspire 2 | up to 5 weeks or until study completion
  Fitbit device track sleep within participants natural environment. The Fitbit Inspire 2 collects data on all stages of sleep throughout night, which helps to calculate sleep efficiency.

CONTACTS AND LOCATIONS:
Locations (1):
- University of the Sciences, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No